





# Über die Rolle von Adjuvantien bei der Stimulierung von angeborenen Immunreaktionen nach Allergen Immuntherapie

Originaltitel der Studie (Englisch):

A Comparison of innate immune responses induced by allergy immunotherapy with different adjuvants

Dieses Forschungsprojekt ist organisiert durch:

- Prof. Dr. sc. nat. Pål Johansen, Dermatologische Klinik, UniversitätsSpital Zürich, Gloriastrasse 31, 8091 Zürich, Schweiz
- Prof Dr. med. Ludger Klimek, Allergiezentrum Wiesbaden, An den Quellen 10, 65183 Wiesbaden, Deutschland

Sehr geehrte Dame, sehr geehrter Herr,

Wir möchten Sie anfragen, ob Sie an einem Forschungsprojekt teilnehmen wollen. Im Folgenden wird Ihnen das geplante Forschungsprojekt dargestellt:

# **Detailliertere Information**

# 1. Ziel des Projekts

Wir wollen mit diesem Projekt untersuchen, ob Immunreaktionen in den ersten Tagen nach Allergen Immuntherapie (AIT) in Blut nachgewiesen können. Dabei soll vor ihrer mit dem Allergologen vereinbarten AIT sowie 1, 7 und 49 Tage danach eine Blutentnahme gemacht werden. Dies würde uns erlauben die Immunreaktionen im Labor zu testen.

### 2. Auswahl

Es können alle Personen teilnehmen, die an einer allergischen Krankheit leiden und/oder für solche behandelt werden. Ausserdem müssen Sie älter als 18 Jahr sein.

# 3. Allgemeine Informationen zum Projekt

Es handelt sich um ein Forschungsprojekt, das im UniversitätsSpital Zürich (CH) in Zusammenarbeit mit dem Allergiezentrum Wiesbaden (DE) durchgeführt wird. An dem Projekt werden 24 Patienten teilnehmen (16 davon in Zürich und 8 in Wiesbaden), die wegen Sensibilisierung auf Gräserpollen oder Birkenpollen an einer allergischen Rhinokonjunktivitis leiden und sich für eine Allergen Immuntherapie in Zürich oder Wiesbaden entschieden haben. Vor der Immuntherapie sowie einen Tag und sieben Tage später wird im Rahmen des Forschungsprojektes eine Blutentnahme gemacht. Bei

Laboruntersuchungen wird das Blut auf entzündliche Zellen (z.B. Leukozyten) und Moleküle (z.B. Enzyme, Zytokine und Antikörper) analysiert. Das Ziel ist es, zu testen wie die verschiedenen in der Immuntherapie enthaltenden Adjuvantien (Immunreaktionsverstärker) die gemessenen Entzündungsreaktionen beeinflussen. Das Forschungsprojekt wird gemäss der in der Schweiz bzw. in Deutschland geltenden Gesetzgebung durchgeführt. Die zuständige Ethikkommission hat dieses Projekt geprüft und bewilligt.

# 4. Ablauf

Wenn Sie bereit sind, an diesem Projekt teilzunehmen, werden Sie von einer Prüfärztin oder einem Prüfarzt über das Projekt aufgeklärt. Falls Sie die Voraussetzungen für eine Teilnahme an dem Projekt erfüllen, wird Ihnen kurz vor Ihrer ersten Immuntherapiesitzung (erste Allergenspritze) eine Blutprobe entnommen. Sie werden dann von der Prüfärztin oder dem Prüfarzt gebeten einen Tag, sowie 7 und ca. 49 (±3) Tage später wieder in die Klinik zu kommen für weitere Blutentnahmen. Die letzte Blutentnahme fällt wahrscheinlich zeitlich mit ihrer zweiten Immuntherapiesitzung (zweite Allergenspritze) zusammen. Es wird total ca. 61 Milliliter (ml) Blut entnommen: jeweils 17 ml an den Tagen 0, 1 und 7, und 10 ml am Tag 49. Bei jeder Blutentnahme werden Sie mit der Prüfärztin oder dem Prüfarzt einen Fragebogen beantworten. Das Ausfüllen des Fragebogens wird jedes Mal ca. 5 Minuten in Anspruch nehmen. Nach der letzten Blutentnahme werden Sie von der Studie entlassen.

### 5. Nutzen

Sie werden selbst keinen persönlichen Nutzen an der Projektteilnahme haben. Viele Forschungsergebnisse sind für individuellen Patienten nicht relevant. Ihre Teilnahme an diesem Projekt könnte Ärzten sowie Forschern helfen neue Kenntnisse über die allergenspezifische Immuntherapie sowie Wirkmechanismen der Behandlungsmethode zu gewinnen.

### 6. Rechte

Ihre Teilnahme an dieser Studie ist freiwillig. Wenn Sie nicht mitmachen oder später Ihre Teilnahme zurückziehen wollen, müssen Sie dies nicht begründen. Ihre medizinische Behandlung/Betreuung ist unabhängig von Ihrem Entscheid gewährleistet. Sie dürfen jederzeit Fragen zur Teilnahme und zum Projekt stellen. Wenden Sie sich dazu bitte an die Person, die am Ende dieser Information genannt ist.

### 7. Pflichten

Als Teilnehmer ist es notwendig, dass Sie (i) sich an die notwendigen Vorgaben und Anforderungen durch die Projektleitung halten, und (ii) pünktlich zu geplanten Visiten erscheinen.

# 8. Risiken

Bei einer Teilnahme an dem Projekt sind Sie nur geringfügigen Risiken ausgesetzt. Bei einer Blutentnahme kann es zu Blutergüssen und in ganz seltenen Fällen zu Infektionen kommen.

# 9. Ergebnisse

Die Prüfärztin oder der Prüfarzt bzw. die Projektleitung wird Sie während des siebentägige Forschungsprojekts über alle neuen Erkenntnisse informieren, die den Nutzen oder Ihre Sicherheit und somit Ihre Einwilligung zur Teilnahme beeinflussen können. Bei Zufallsbefunden, die bei Ihnen zur Verhinderung, Feststellung oder Behandlung

bestehender oder künftig zu erwartender Krankheiten beitragen können, werden Sie informiert. Da im Rahmen dieser Forschungsstudie keine medikamentöse oder operative Behandlung gemacht wird, sondern nur Blutentnahmen, werden keine Ergebnisse während des siebentägige Forschungsprojekts vorliegen. Die Ergebnisse der Analysen werden erst nach ihrer Entlassung von der Studie vorliegen. Wenn Sie nicht informiert werden wollen, sprechen Sie bitte mit Ihrem Prüfarzt/der Projektleitung.

# 10. Vertraulichkeit von Daten und Proben

Für dieses Projekt werden Ihre persönlichen und medizinischen Daten erfasst. Nur sehr wenige Fachpersonen werden Ihre unverschlüsselten Daten sehen, und zwar ausschliesslich, um Aufgaben im Rahmen des Projekts zu erfüllen. Bei der Datenerhebung zu Studienzwecken werden die Daten verschlüsselt. Verschlüsselung bedeutet, dass alle Bezugsdaten, die Sie identifizieren könnten (Name, Geburtsdatum), gelöscht und durch einen Schlüssel ersetzt werden. Die Schlüssel-Liste bleibt immer in der Institution (UniversitätsSpital Zürich oder Allergiezentrum Wiesbaden). Diejenigen Personen, die den Schlüssel nicht kennen, können daher keine Rückschlüsse auf Ihre Person ziehen. Bei einer Publikation sind die zusammengefassten Daten daher auch nicht auf Sie als Einzelperson zurückzuverfolgen. Ihr Name taucht niemals im Internet oder einer Publikation auf. Manchmal gibt es die Vorgabe bei einer Zeitschrift zur Publikation, dass Einzel-Daten (sogenannte Roh-Daten) übermittelt werden müssen. Wenn Einzel-Daten übermittelt werden müssen, dann sind die Daten immer verschlüsselt und somit ebenfalls nicht zu Ihnen als Person zurückzuverfolgen. Alle Personen, die im Rahmen des Projekts Einsicht in Ihre Daten haben, unterliegen der Schweigepflicht. Die Vorgaben des Datenschutzes werden eingehalten und Sie als teilnehmende Person haben jederzeit das Recht auf Einsicht in Ihre Daten.

Wenn Daten/ Proben vor Ort gelagert werden, handelt es sich um eine Datenbank/ Biobank für Forschungszwecke.

Probenversand zu anderen Forschungsinstitutionen in der Schweiz oder ins Ausland ist nicht geplant. Sollten die Daten und Proben zur weiterer projektspezifischen Untersuchung weiterversandt werden, werden die vorher verschlüsselt und nur dann versandt. Das Zugriffsrecht auf diese Verschlüsselung hat nur der Leiter dieses Projekts. Verantwortlich für die Einhaltung der nationalen und internationalen Richtlinien zum Datenschutz ist die Projektleitung, die/der im Ausland einen gleichwertigen Datenschutz gewährleistet.

Möglicherweise wird dieses Projekt durch die zuständige Ethikkommission oder durch die Institution, die das Projekt veranlasst hat, überprüft. Der Projektleiter muss eventuell Ihre persönlichen und medizinischen Daten für solche Kontrollen offenlegen.

Es ist möglich, dass Ihr nachbehandelnder Arzt kontaktiert wird, um Auskunft über Ihren Gesundheitszustand zu geben.

# 11. Behördliche Einsicht in der Studie

Die Projektleitung wird bei Anfragen der Ethikkommission oder anderen Gesundheits- oder Aufsichtsbehörden direkte Zugriff und Einsicht auf die ursprünglichen medizinischen Unterlagen des Probanden gewährt, um Projektvorgehen oder Daten zu überprüfen. Dieser Zugriff wird gewährt ohne ihre Vertraulichkeit zu verletzen.

### 12. Rücktritt

Die Teilnahme in diesem Forschungsprojekt basiert auf Freiwilligkeit. Sie können jederzeit Ihre Teilnahme beenden und von dem Projekt zurücktreten, wenn Sie dies wünschen. Die bis dahin erhobenen Daten und Proben werden noch verschlüsselt ausgewertet, da das ganze Projekt sonst seinen Wert verliert.

Es ist nicht möglich, Ihre Daten und Proben bei Rücktritt zu anonymisieren, d.h. die Daten und Proben bleiben weiterhin verschlüsselt. Prüfen Sie bitte, ob Sie damit einverstanden sind, bevor Sie bei dem Projekt mitmachen.

# 13. Entschädigung

Wenn Sie an diesem Projekt teilnehmen, bekommen Sie dafür keine Entschädigung. Wenn sie Reisekosten in Zusammenhang mit der Studie haben, werden diese von der Projektleitung entschädigt.

# 14. Haftung

- A) USZ: Falls Sie durch die Studie einen gesundheitlichen Schaden erleiden, haftet das UniversitätsSpital Zürich ("Versicherung für Klinische Versuche und Nicht Klinische Versuche", Zürich Versicherungsgesellschaft AG, Policenummer 14.970.888)
- B) AZW: Für Patienten die das AZW besuchen, gilt bei einem gesundheitlichen Schaden die dortige Patientenversicherung wie es im Bewilligung an Prof. Klimek der Mannheimer Ethikkommission gehalten ist.

# 15. Finanzierung

Das Projekt wird von Forschungsgeldern der Universität Zürich finanziert.

# 16. Kontaktperson(en)

Bei allen Unklarheiten, Befürchtungen oder Notfällen, die während des Projekts oder danach auftreten, können Sie sich jederzeit an eine dieser Kontaktpersonen wenden.

# **UniversitätsSpital Zürich:**

Prof. Dr. sc. nat. Pål Johansen (Leiter)

Email pal.johansen@usz.ch

Tel +41 (0)44 255 8616

Dr. med. Deborah Leuthard (Prüfärztin)

Email deborah.leuthard@usz.ch

Tel +41 (0)43 253 0568

Dr. med. Sara Micaletto (Allergologin)

Email sara.micaletto@usz.ch

Tel +41 (0)43 253 7630

Dr. med Eugen Bersuch (Allergologe)

Email: <a href="mailto:eugen.bersuch@usz.ch">eugen.bersuch@usz.ch</a>

Tel +41 (0)43 253 8580

Frau Elvira Schmid (Pflegeleiterin der

Allergiestation)

Email elvira.schmid@usz.ch

Tel +41 (0)44 255 2441

**Notfall USZ:** Tel +41 (0)44 255 11 11

Allergiezentrum Wiesbaden:

Prof. Dr. med. Ludger Klimek (Leiter)

Email: ludger.klimek@allergiezentrum.org

Tel: +49 (0)611 308 608-0

Dr. med. Annette Sperl (Allergologin)

Email: annette.sperl@allergiezentrum.org

Tel: +49 (0)611 308 608-0

Cand. med. Alina Müller (Prüfärztin)

Email: <u>alina.mueller@usz.ch</u>

Tel: +41 (0)76 391 18 35

Dr. Ingrid Casper (Studiekoordinatorin)

Email ingrid.casper@allergiezentrum.org

Tel +49 (0)611 308 608-257







# Schriftliche Einverständniserklärung des Patienten zur Teilnahme an einer Forschungsstudie

- Bitte lesen Sie dieses Formular sorgfältig durch.
- Bitte fragen Sie, wenn Sie etwas nicht verstehen oder wissen möchten

### **BASEC-Nummer: 2019-01233**

# Nummer der Studie USZ-AZW\_MCT001

**Titel der Studie** A Comparison of innate immune responses induced by allergy immunotherapy with different adjuvants

**Sponsor** Dermatologische Klinik, UniversitätsSpital Zürich & Universität Zürich, Gloriastrasse 31, 8091 Zürich, Schweiz

Ort der Studie UniversitätsSpital Zürich (CH) und Allergiezentrum Wiesbaden (DE)

**Leiter/Leiterin des Projekts:** Prof. Dr. sc. nat. Pål Johansen (USZ), Prof. Dr. med. Ludger Klimek (AZW)

**Prüfarzt/ Prüfperson** Dr. med. Deborah Leuthard (USZ) und Dr. med. Annette Sperl (AZW), med. pract. Alina Müller (USZ/AZW)

# Patientin/Patient

Name und Vorname Geburtsdatum Geschlecht

männlich / weiblich

- Ich wurde vom unterzeichnenden Arzt mündlich und schriftlich über die Ziele und den Ablauf der Studie USZ-AZW\_MCT001, über die zu erwartenden Wirkungen, über mögliche Vor- und Nachteile sowie über eventuelle Risiken informiert.
- Ich habe die zur oben genannten Studie abgegebene schriftliche Patienteninformation vom 9. August 2019 gelesen und verstanden. Meine Fragen im Zusammenhang mit der Teilnahme an dieser Studie sind mir zufriedenstellend beantwortet worden. Ich kann die schriftliche Patienteninformation behalten und erhalte eine Kopie meiner schriftlichen Einverständniserklärung.
- Ich hatte genügend Zeit, um meine Entscheidung zu treffen.
- Ich bin darüber informiert, dass eine Versicherung Schäden deckt, falls solche im Rahmen der Studie auftreten.
- Ich weiss, dass meine Daten und Proben nur in verschlüsselter Form im Rahmen dieser Studie weitergegen werden können.

- Ich bin einverstanden, dass die zuständigen Fachleute des Studienauftraggebers, der Behörden und der Kantonalen Ethikkommission zu Prüf- und Kontrollzwecken in meine Originaldaten Einsicht nehmen dürfen, jedoch unter strikter Einhaltung der Vertraulichkeit.
- Ich nehme an dieser Studie freiwillig teil. Ich kann jederzeit und ohne Angabe von Gründen meine Zustimmung zur Teilnahme widerrufen, ohne dass mir deswegen Nachteile bei der weiteren medizinischen Betreuung entstehen. In diesem Fall werde ich zu meiner Sicherheit abschliessend medizinisch untersucht.
- Ich bin mir bewusst, dass während der Studie die in der Patienteninformation genannten Anforderungen und Einschränkungen einzuhalten sind. Im Interesse meiner Gesundheit kann mich der Prüfarzt jederzeit von der Studie ausschliessen.

| Ort, Datum | Unterschrift der Patientin/des Patienten |
|------------|------------------------------------------|
| | · |

**Bestätigung des Prüfarztes/ der Prüfperson:** Hiermit bestätige ich, dass ich diesem Patienten/dieser Patientin Wesen, Bedeutung und Tragweite der Studie erläutert habe. Ich versichere, alle im Zusammenhang mit dieser Studie stehenden Verpflichtungen zu erfüllen. Sollte ich zu irgendeinem Zeitpunkt während der Durchführung der Studie von Aspekten erfahren, welche die Bereitschaft des Patienten/der Patientin zur Teilnahme an der Studie beeinflussen könnten, werde ich ihn/sie umgehend darüber informieren.

Ort, Datum Unterschrift des Prüfarztes/ der Prüfperson